CLINICAL TRIAL: NCT00437918
Title: Phase IV Study on Predictive Markers for the Effectiveness of Nateglinide or Acarbose for Controlling Post-Prandial Glucose in Type 2 Diabetics Already on Optimized Insulin Glargine Therapy
Brief Title: The Effects of Nateglinide and Acarbose on the Post-Prandial Glucose Control in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inje University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Jeong Hyun Park, MD PhD / Professor, Inje University Pusan Paik Hospital / Paik Diabetes Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDC-07-01
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Nateglinide; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: nateglinide
Drug: acarbose

SUMMARY:
In type 2 diabetic patients, tight blood glucose control often requires both fasting and post-prandial glucose control separately. In the diabetic patients already on the insulin glargine treatment for the control of fasting blood glucose, additional measures for the control of post-prandial glucose level are often required. Nateglinide and acarbose are frequently used for this purpose. We hypothesized that the short acting sulfonylurea "nateglinide" may be more efficacious in diabetic patients with appreciable endogenous insulin secretion, while acarbose may be more efficacious in patients with lower endogenous insulin secretion. And we also want to clarify the clinical and biochemical parameters that can predict the responsiveness to each agent in this multi-center randomized open cross-over clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Korean
* Type 2 diabetes mellitus
* No prior history of diabetic ketoacidosis
* HbA1c between 7.5-10.0%

Exclusion Criteria:

* Type 1 diabetes mellitus
* Gestational diabetes mellitus
* Secondary diabetes mellitus
* Severe hyperglycemia with symptoms
* Severe chronic diabetic complications (PDR,s-Cr>1.3mg/dL)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
7 point SMBG (self monitoring of blood glucose)

SECONDARY OUTCOMES:
HOMA-beta for predicting the effectiveness of each agents

CONTACTS AND LOCATIONS:
Overall Officials: Jeonghyun Park, MD PhD, Principal Investigator — Director, Paik Diabetes Center, Pusan Paik Hospital, College of Medicine, Inje University
Locations (2):
- South Korea (2):
  - Paik Diabetes Center, Pusan Paik Hospital, College of Medicine, Inje University, Busan
  - Endocrinology and Metabolism, Maryknoll General Hospital, Busan

REFERENCES:
- [Derived] Kim MK, Suk JH, Kwon MJ, Chung HS, Yoon CS, Jun HJ, Ko JH, Kim TK, Lee SH, Oh MK, Rhee BD, Park JH. Nateglinide and acarbose for postprandial glucose control after optimizing fasting glucose with insulin glargine in patients with type 2 diabetes. Diabetes Res Clin Pract. 2011 Jun;92(3):322-8. doi: 10.1016/j.diabres.2011.01.022. Epub 2011 Mar 3. PMID 21376417